CLINICAL TRIAL: NCT05934097
Title: A Phase 1b, Open-Label, Multicenter Study of FT596 in Combination With R-CHOP in Subjects With B-Cell Lymphoma
Brief Title: FT596 in Combination With R-CHOP in Subjects With B-Cell Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was withdrawn (Sponsor decision).
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FT596-102
Record Dates: First submitted 2023-04-30; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Diffuse Large B Cell Lymphoma; Transformed Indolent Non-Hodgkin's Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to one of 2 treatment regimens corresponding to different schedules (standard or alternate) of R-CHOP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A (FT596 in combination with standard schedule R-CHOP) (Experimental): FT596 in combination with standard schedule R-CHOP (rituximab, cyclophosphamide, doxorubicin, and vincristine on Day 1; prednisone on Days 1-5; and FT596 on Day 8) for a total of six 21-day cycles.
  Interventions: Drug: FT596; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Rituximab; Drug: Bendamustine
- Regimen B (FT596 in combination with alternate schedule R-CHOP) (Experimental): FT596 in combination with alternate schedule R-CHOP (prednisone on Days 1-5; rituximab, cyclophosphamide, doxorubicin, and vincristine on Day 5; and FT596 on Day 8) for a total of six 21-day cycles
  Interventions: Drug: FT596; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Rituximab; Drug: Bendamustine

INTERVENTIONS:
Drug: FT596 — Dosing to be initiated at a dose no higher than highest tolerable dose in study FT596-101, intravenously
Drug: Cyclophosphamide — 750 mg/m^2 intravenously
Drug: Doxorubicin — 50 mg/m^2 intravenously
Drug: Vincristine — 1.4 mg/m^2 (maximum dose 2 mg) intravenously
Drug: Prednisone — 100 mg orally
Drug: Rituximab — 375 mg/m^2 intravenously
  Other Names: Rituxan; Truxima; Ruxience
Drug: Bendamustine — 90 mg/m^2 IV infusion
  Other Names: Bendeka; Treanda

SUMMARY:
This is a Phase I study of FT596 in combination with two different schedules (standard or alternate) of R-CHOP in subjects with B-cell lymphoma who are previously untreated or have received no more than one prior line of treatment. The study will consist of a dose-escalation stage followed by a dose-expansion stage.

DETAILED DESCRIPTION:
This is a Phase I study of FT596 in combination with 2 different schedules (standard or alternate) of R-CHOP in subjects with B-cell lymphoma who are previously untreated or have received no more than one prior line of treatment.

The study will evaluate both the clinical benefit of FT596 when combined with R-CHOP given on a standard or alternate schedule.

Subjects will be enrolled in two stages: a dose-escalation stage and a dose-expansion stage. After safety and tolerability have been assessed to define the maximum tolerated dose (MTD) (or the maximum assessed dose [MAD] in the absence of dose limiting toxicities [DLTs] defining the MTD) in the dose-escalation stage, the dose-expansion stage will further evaluate the safety and activity of FT596 in combination.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of B-cell lymphoma (BCL) as described below:

  * Histologically documented BCL
  * Previously untreated or no more than one prior systemic therapy for BCL
  * At least one bi-dimensionally measurable lesion
  * Subjects with >1 measurable lesion agreement to undergo a biopsy
* Capable of giving signed informed consent
* Age ≥ 18 years old
* Stated willingness to comply with study procedures through study duration
* Contraception use for women and men as defined in the protocol
* Negative serum pregnancy test within 7 days of treatment for women

Key Exclusion Criteria:

* Prior anthracycline therapy
* Females who are pregnant or breastfeeding
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥2
* Evidence of insufficient organ function
* Currently receiving or likely to receive systemic immunosuppressive therapy
* Receipt of allograft organ transplant
* Known active central nervous system (CNS) involvement by malignancy
* Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Clinically significant cardiovascular disease
* Positive HIV test
* Positive Hepatitis B (HBV) or Hepatitis C (HCV) test
* Live vaccine <6 weeks prior to start of conditioning
* Allergy to human albumin or dimethyl sulfoxide (DMSO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2039-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities within each dose escalation cohort | Day 21
Nature of dose-limiting toxicities within each dose escalation cohort | Day 21
Incidence, nature, and severity of adverse events (AEs) of FT596 in combination with R-CHOP in B-cell lymphoma previously untreated or no more than one previous line of therapy with severity determined according to NCI CTCAE, v5.0 | Up to 5 years

SECONDARY OUTCOMES:
Investigator-assessed complete response (CR) | Up to 2 years
  Proportion of subjects who achieve a complete response (CR) per Lugano 2014 classification
Investigator-assessed objective-response rate (ORR) | Up to 2 years
  Proportion of subjects who achieve a partial response (PR) or complete response (CR) per Lugano 2014 classification
Investigator-assessed duration of response (DOR) | Up to 15 years
  Duration from the first occurrence of a documented objective response until the time of disease progression or relapse, or death from any cause, whichever occurs first, per Lugano 2014 classification
Investigator-assessed duration of complete response (DoCR) | Up to 15 years
  Duration from the first occurrence of a documented complete response (CR), per Lugano 2014 classification until the time of disease progression or relapse, or death from any cause, whichever occurs first
Progression-free survival (PFS) | Up to 15 years
  Time from first dose of study treatment to progressive disease (PD), or to the day of death for any reason, whichever occurs earlier, based on Lugano 2014 classification
Overall survival (OS) | Up to 15 years
  Time from first dose of study treatment to death from any cause
Area Under the Plasma Concentration Time Curve (AUC) of FT596 | Cycles 1-6 (each cycle is 28 days): Days 1,8,11,15,18; and Post-Treatment Week 1, Week 2, Week 4, and Week 8
  Assessed by the detection of FT596 in peripheral blood following FT596 administration.
Maximum Plasma Concentration (Cmax) of FT596 | Cycles 1-6 (each cycle is 28 days): Days 1,8,11,15,18; and Post-Treatment Week 1, Week 2, Week 4, and Week 8
  Assessed by the detection of FT596 in peripheral blood following FT596 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Fate Trial Disclosure, Study Director — Fate Therapeutics

IPD SHARING:
Plan to Share IPD: No